CLINICAL TRIAL: NCT01100203
Title: Aldosterone Blockade in Chronic Kidney Disease. Influence on Arterial Stiffness and Kidney Function
Brief Title: Aldosterone Blockade in Chronic Kidney Disease: Influence on Arterial Stiffness and Kidney Function
Acronym: ALBLOCK-2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: It was not possible within the time frame to recruit the planned no. of patients.
Sponsor: Lene Boesby (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor-Investigator, Lene Boesby, MD, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALBLOCK-2
Record Dates: First submitted 2010-04-06; First posted 2010-04-08 (Estimated); Last update posted 2012-02-08 (Estimated); Status verified 2012-02

CONDITIONS: Chronic Kidney Disease
Keywords: aldosterone receptor inhibition; arterial stiffness; ambulatory arterial stiffness index
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Eplerenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Active Comparator)
  Interventions: Drug: Eplerenone
- Control (No Intervention)

INTERVENTIONS:
Drug: Eplerenone — 25 mg once daily 1 week, then 50 mg once daily for another 23 weeks.
  Arms: Treatment

SUMMARY:
Patients with Chronic Kidney Disease (CKD) have a poor prognosis primarily due to cardiovascular disease. The cardiovascular risk can be assessed by measurements of arterial stiffness. A decrease in stiffness has been shown to decrease the risk of cardiovascular disease as well as death. Most of the CKD population also have hypertension and the control of blood pressure is one of the corner stones in inhibition of disease progression. Using drugs that specifically block the renin-angiotensin-system for blood pressure control has been shown to have a beneficial impact on inhibition of progression beyond that of the achieved blood pressure control. It has been reported that inhibition of the hormone aldosterone has a positive effect on survival in patients with heart failure, hypertension and diabetic as well as on-diabetic nephropathy.

This study undertakes the investigation of the influence on arterial stiffness of adding an aldosterone receptor inhibitor to the medication CKD patients are already taking. Besides the primary end point which is Pulse wave velocity (PWV), arterial stiffness is also quantified thorough ambulatory blood pressure measurements.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years age ≤ 80 years age
* voluntarily signed informed consent
* 15 ml/min/1,73 m2 ≤ estimated Glomerular Filtration Rate < 60 ml/min/1,73 m2
* BP ≥ 130/80 mmHg or undergoing anti-hypertensive treatment

Exclusion Criteria:

* p-potassium is > 5.0 mM
* allergy to contents
* treated with spironolactone
* treated with potent inhibitors of CYP3A4 (see SPC for details)
* treated with lithium, ciclosporin, tacrolimus, prednisolone, or other immunosuppressing drug
* inborn errors of metabolism (see SPC for details)
* pregnancy or lactation
* fertile woman, not using safe contraception devices
* dementia or other psychiatric disorder, making understanding of the study conditions impossible
* other severe, chronic illness besides CKD, including liver insufficiency, according to investigators' judgement
* vascular surgery including stenting or graft implantation on a. brachialis, aorta or the carotid arteries
* systolic BP > 200 mmHg
* immeasurable pulse amplitude

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2010-04; Primary Completion 2012-01 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Pulse wave velocity | 24 weeks
  Pulse wave velocity measured using the SphygmoCor device.
Pulse Wave velocity | 12 weeks
Pulse wave velocity | baseline

SECONDARY OUTCOMES:
Ambulatory arterial stiffness index | 24 weeks
  24 hour ambulatory blood pressure measurements, give rise to the index, which is a secondary measure of arterial compliance.
Pulse wave analysis | 24 weeks
  Parameters are Augmentation Index, subendocardial viability ratio, pulse, time to reflection, ejection duration.
Albuminuria | baseline
  Will be calculated from 24 hour urine collections.
Pulse wave analysis | baseline
Ambulatory arterial stiffness index | baseline
Ambulatory arterial stiffness index | 12 weeks
Pulse wave analysis | 12 weeks
Albuminuria | 12 weeks
Albuminuria | 24 weeks
Estimated glomerular filtration rate (eGFR) | baseline
  Estimated glomerular filtration rate (eGFR) will be calculated by using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula.
Estimated glomerular filtration rate (eGFR) | 12 weeks
Estimated glomerular filtration rate (eGFR) | 24 weeks
Plasma potassium | baseline
Plasma potassium | week 1
Plasma potassium | week 2
Plasma potassium | week 4
Plasma potassium | week 8
Plasma potassium | week 12
Plasma potassium | week 16
plasma potassium | week 20
plasma potassium | week 24
Blood pressure | baseline
  BP will be measured at all visits
Blood pressure | 12 weeks
Blood pressure | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lene Boesby, MD, Principal Investigator — Herlev Hospital
Locations (2):
- Denmark (2):
  - Dept. Nephrology, Herlev Hospital, Herlev
  - Herlev Hospital, Herlev

REFERENCES:
- [Derived] Chung EY, Ruospo M, Natale P, Bolignano D, Navaneethan SD, Palmer SC, Strippoli GF. Aldosterone antagonists in addition to renin angiotensin system antagonists for preventing the progression of chronic kidney disease. Cochrane Database Syst Rev. 2020 Oct 27;10(10):CD007004. doi: 10.1002/14651858.CD007004.pub4. PMID 33107592
- [Derived] Boesby L, Elung-Jensen T, Strandgaard S, Kamper AL. Eplerenone attenuates pulse wave reflection in chronic kidney disease stage 3-4--a randomized controlled study. PLoS One. 2013 May 21;8(5):e64549. doi: 10.1371/journal.pone.0064549. Print 2013. PMID 23704994